CLINICAL TRIAL: NCT02211664
Title: Physician-Initiated Trial Investigating the Efficacy of Endovascular Treatment of Femoropopliteal Arterial Stenotic Disease With the Biotronik Passeo-18 Lux Drug Releasing Balloon and the Biotronik Pulsar-18 Stent (Comparing With 4EVER Trial Results)
Acronym: BIOLUX 4EVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-120130
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

ARMS (1):
- Passeo-18-Lux & Pulsar-18 (Experimental): The interventional procedure sequence consists of the following steps:
  1. pre-dilation of the lesion with a Passeo-18 balloon (mandatory)
  2. dilation of the lesion with a Passeo-18 Lux drug releasing balloon (mandatory); a maximum of 2 Passeo-18 Lux balloons can be used per lesion (drug load cannot exceed 12µg)
  3. stenting of the lesion with a Pulsar-18 stent (mandatory)
  4. post-dilation of the lesion with a Passeo-18 balloon (not mandatory)
  Interventions: Device: Passeo-18 balloon; Device: Passeo-18 Lux drug releasing balloon; Device: Pulsar-18 stent

INTERVENTIONS:
Device: Passeo-18 balloon
Device: Passeo-18 Lux drug releasing balloon
Device: Pulsar-18 stent

SUMMARY:
The objective of this clinical investigation is to evaluate the short- and long-term (up to 24 months) outcome of treatment by means of dilation with the Passeo-18 Lux drug releasing balloon and by Pulsar-18 stent implantation in symptomatic (Rutherford 2-4) femoro-popliteal arterial stenotic or occlusive lesions.

DETAILED DESCRIPTION:
Ever since its introduction, one of the major limitations of endovascular therapy is the occurrence of restenosis after treatment. Factors contributing to loss of primary patency after percutaneous transluminal angioplasty (PTA) due to balloon injury are negative arterial remodeling, excessive neointimal proliferation and elastic recoil. In order to increase sustained vessel patency, systemic medication administration and brachytherapy have been proposed, but have not led to any success. With the introduction of stents, patency rates have been optimized also on longer term. However, neointimal hyperplasia after endovascular stent placement in infra-inguinal arteries remains a major limiting issue. Stents themselves contribute to this excessive intimal formation because of the vascular response to the metallic prosthesis. In order to find a solution to overcome this limitation, the possibilities of drug-eluting technologies are being examined.

Current concepts include drug-eluting stents (DES), which provide sustained release of anti-proliferative medication into the vessel wall. The application of a drug coating on a stent surface inhibits the inflammatory response and smooth muscle cell proliferation in the vessel wall during a certain period and delays the process of intimal hyperplasia. Thus, DES technology was developed to prevent early restenosis and late luminal loss to potentially improve long-term patency rates. Because DES with active stent coatings have shown to be beneficial in the treatment of coronary artery disease, the technique of active stent coatings (sirolimus or paclitaxel) as commonly used in coronary interventions was transferred to the infrainguinal vascular bed. However, an active stent coating (sirolimus or paclitaxel) only inhibits the inflammatory response and smooth muscle cell proliferation in the vessel wall for a certain period; in fact, it merely delays the process of intimal hyperplasia as demonstrated by the 2-year results of the SIROCCO study.

Another novel way of inhibiting restenosis after PTA is the use of drug-coated balloons (DCB), which inhibit restenosis by an immediate local release of medication during the intervention. The rationale behind the use of DCBs is based on the finding that sustained drug elution is not a necessary to obtain a sustained inhibition of restenosis. The concept of using a balloon with medication to treat vascular disease was introduced in 2003 by Scheller et al.

One of the most commonly used drugs for arterial applications is the anti-proliferative paclitaxel (Taxol), which impedes cell division in the cell cycle. Paclitaxel has certain characteristics which make it a promising candidate for treatment of peripheral arterial disease. Because it is hydrophobic, paclitaxel does not require the use of a polymer to prevent wash-off during tracking or implantation. Adequate drug delivery to the vessel wall is possible because of its lipophilic characteristic, which enables paclitaxel to interact with the high concentrations of lipids present in the vessel wall and avoids the need for a polymer. Results of preclinical and clinical studies have shown that short-term exposure to Paclitaxel may suffice to obtain a sustained reduction in late lumen loss and avoid restenosis in both coronary and peripheral arteries: in contrast to stents, DCBs do not leave any residual material in the artery lumen that could trigger neointimal proliferation, thus making DCBs an attractive alternative to stents, especially in challenging arterial anatomies. Further investigation is warranted in order to obtain conclusive data. Furthermore, the benefit of treating in-stent restenosis (ISR) in the peripheral arteries with DCBs has yet to be investigated, although limited data is already available to date.

The clinical value of these drug-eluting technologies has been proven repeatedly in the coronary arteries, and evidence of therapeutic applications to peripheral artery disease is starting to build. It is the intent of this prospective study to evaluate the treatment of a drug-coated balloon followed by stent implant and comparing this to the results of the 4EVER trial and results in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. General Inclusion Criteria:

   * De novo lesions located in the femoropopliteal arteries suitable for endovascular treatment
   * Patient presenting with a score from 2 to 4 according to the Rutherford classification
   * Patient is willing to comply with specified follow-up evaluations at the predefined time intervals time
   * Patients is >18 years old
   * Patient understands the nature of the procedure and provides written informed consent, prior to enrollment in the study
   * Prior to enrollment, the target lesion was crossed with standard guidewire manipulation
2. Angiographic Inclusion Criteria:

   * The target lesions are located within the native SFA: distal point 3 cm above knee joint and 1 cm below the origin of the profunda femoralis
   * The target lesion has angiographic evidence of stenosis >50% or occlusion
   * Length of the target lesion is ≤ 19 cm by visual estimation and can be covered with one stent
   * Target vessel diameter visually estimated is ≥4 mm and ≤6 mm
   * There is angiographic evidence of at least one-vessel-runoff to the foot

Exclusion Criteria:

* Presence of another stent in the target vessel that was placed during a previous procedure
* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
* Previous bypass surgery in the same limb
* Patients contraindicated for antiplatelet therapy, anticoagulants or thrombolytics
* Patients who exhibit persistent acute intraluminal thrombus at the target lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than 12 months
* Ipsilateral iliac artery treatment before target lesion treatment with a residual stenosis > 30%
* Use of thrombectomy, atherectomy or laser devices during procedure
* Any planned surgical intervention/procedure 30 days after the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not reached the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months | 12 months
  Defined as freedom from >50% restenosis as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no reintervention.

SECONDARY OUTCOMES:
Technical success | 1 day post-op
  Defined as the ability to cross and stent the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex imaging.
Procedural success | 1 day post-op
  Defined as the ability to perform the procedure as stated in the protocol, with the Biotronik portfolio.
Number of puncture site complications | 1 day post-op
Compression time | 1 day post-op
  In patients when manual compression is applied to close the puncture site (instead of a closure device).
Primary patency rate at 1-month follow-up | 1 month
  Defined as freedom from >50% restenosis as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no re-intervention.
Primary patency rate at 6- and 24-month follow-up | 6 and 24 months
  Defined as freedom from >50% restenosis as indicated on a duplex ultrasound with peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no re-intervention.
Freedom from Target Lesion Revascularization (TLR) at at 1-, 6-, 12- and 24-months follow-up | 1, 6, 12 and 24 months
  Defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal an distal to the treated lesion edge.
Clinical success at 1-, 6-, 12- and 24-months follow-up | 1, 6, 12, 24 months
  Defined as an improvement of Rutherford classification at 1-, 6-, 12- and 24-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Changes in ABI measurements at 1-, 6-, 12- and 24-months | 1, 6, 12, 24 months
  Defined as the ankle-brachial index (ABI) measurement difference at 1-, 6-, 12- and 24-months compared to the pre-procedure ABI measurement.
Serious Adverse Events | up to 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - University Hospital Antwerp, Edegem, Antwerp
  - OLV Hospital, Aalst
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - RZ Heilig Hart Hospital, Tienen

REFERENCES:
- [Derived] Deloose K, Bosiers M, Peeters P, Verbist J, Maene L, Beelen R, Keirse K, Hendriks J, Lauwers P, Wauters J, Verschueren M. Combining the Passeo-18 Lux Drug-Coated Balloon and the Pulsar-18 Bare Metal Stent: 12- and 24-Month Outcomes of the BIOLUX 4EVER Investigator-Initiated Trial. J Endovasc Ther. 2020 Dec;27(6):936-945. doi: 10.1177/1526602820952413. Epub 2020 Sep 1. PMID 32873131